CLINICAL TRIAL: NCT00361075
Title: Mentored Patient Oriented Research Career Development Award
Brief Title: Midlife Cholesterol Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Washington (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 5K23RR016067-05 (NIH)
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Menopause; Postmenopause; Premenopause; Cardiovascular Disease
Keywords: Perimenopause; Abdominal adipose tissue; Women's health; Cholesterol; Lipid Metabolism
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Estradiol; Estrogens; Progesterone

INTERVENTIONS:
Drug: transdermal estradiol patch (Vivelle), oral estrogen (Estrace), progesterone (Prometrium)

SUMMARY:
The postmenopausal state is associated with an increase risk for heart disease. Much of this increase in risk may be due to the loss of estrogen (the main female hormone) and the effect of this loss on lipids (blood fats). This loss of estrogen is often treated by estrogen replacement therapy. Estrogen replacement therapy seems to have a beneficial effect on lipid levels. The purpose of this research study is to understand 1) how menopause affects lipids and 2) how hormone replacement therapy effects the lipid metabolism of postmenopausal women.

DETAILED DESCRIPTION:
Women with the Metabolic Syndrome (central obesity, insulin resistance, and dyslipidemia) are at especially high risk for coronary heart disease (CHD). The prevalence of the Metabolic Syndrome increases with menopause and may partially explain the acceleration in CHD after menopause. Menopause is associated with increased central adiposity, insulin resistance, dyslipidemia (hypertriglyceridemia, increased low density lipoprotein (LDL), reduced high density lipoprotein (HDL) and small dense LDL particles), and increased thrombotic/inflammatory states, but there are no studies investigating the mechanisms that mediate these changes. The objectives of the proposed project are to investigate the emergence of the features of the Metabolic Syndrome in women followed prospectively through the menopause and determine if these features can be reversed with transdermal estrogen. We hypothesize that the increase in central adiposity with menopause will be a major contributor to the increased prevalence of the Metabolic Syndrome with menopause. This is the first prospective study to investigate the 1) effects of menopause and 2) estrogen replacement therapy (ERT) (oral vs. transdermal) on features of the Metabolic Syndrome. We will determine if the increase in central (intraabdominal)fat with menopause is associated with changes in lipids, insulin resistance, adipocytokines, and fibrinolytic/inflammatory markers. We will then determine if these changes can be reversed with transdermal ERT, as compared to oral ERT, which has pharmacologic effects on the liver.

ELIGIBILITY:
Inclusion Criteria:

* Have demonstrated an interest to participate in the ERT trial
* Be premenopausal (have menstrual period in previous three months) prior to start of observational arm
* Prior to start of interventional arm (ERT), the women must be postmenopausal (have not had a menstrual cycle in the past twelve months and FSH >30)
* Be between the ages of 47 and 55
* Not be taking any form of estrogen replacement
* Have an intact uterus and at least one ovary and normal screening mammogram in the 12 months prior to starting ERT

Exclusion Criteria:

* Body mass index (kg/m2) greater than 40 kg/m2
* History of diabetes mellitus or fasting >110 mg/dl at screening
* Abnormal fasting LDL or triglyceride
* Use of lipid lowering medications, beta-blockers, birth control pills
* Active liver disease (recent history of active hepatitis, jaundice, scleral icterus, and/or elevated liver function tests
* History of breast, endometrial or ovarian cancer
* History of thrombotic disorder (past history of pulmonary embolus or deep venous thrombosis) or known history of CAD

Ages: 47 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120
Dates: Start 1998-07; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
LDL particle size and density

SECONDARY OUTCOMES:
Total body adiposity (Dexa scans)
Intra-abdominal fat (CT scans)
Lipid Profile
Inflammatory Factors
Adipocytokines

CONTACTS AND LOCATIONS:
Overall Officials: Molly C. Carr, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Carr MC, Hokanson JE, Deeb SS, Purnell JQ, Mitchell ES, Brunzell JD. A hepatic lipase gene promoter polymorphism attenuates the increase in hepatic lipase activity with increasing intra-abdominal fat in women. Arterioscler Thromb Vasc Biol. 1999 Nov;19(11):2701-7. doi: 10.1161/01.atv.19.11.2701. PMID 10559014
- [Background] Carr MC, Kim KH, Zambon A, Mitchell ES, Woods NF, Casazza CP, Purnell JQ, Hokanson JE, Brunzell JD, Schwartz RS. Changes in LDL density across the menopausal transition. J Investig Med. 2000 Jul;48(4):245-50. PMID 10916282